CLINICAL TRIAL: NCT03943927
Title: Preemptive Pharmacogenetic- Guided Metoprolol Management for Postoperative Atrial Fibrillation in Cardiac Surgery: The PREEMPTIVE- Pilot Trial
Brief Title: Preemptive Pharmacogenetic-guided Metoprolol Management for PostoperativeAtrial Fibrillation in Cardiac Surgery
Acronym: PREEMPTIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Miklos Kertai, Professor of Anesthesiology, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 190578
Record Dates: First submitted 2019-05-07; First posted 2019-05-09 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Post-operative Atrial Fibrillation
Keywords: Metoprolol; Genotype; Phenotype; CYP2D6

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pharmacogenetic-guided metoprolol management (Experimental)
  Interventions: Other: Guided Metoprolol Management

INTERVENTIONS:
Other: Guided Metoprolol Management — CYP2D6 Genotyping: Consented patients will have blood drawn for genotyping prior to surgery. Patients will be classified as poor metabolizers, intermediate metabolizers, extensive (normal) metabolizers, or ultrafast metabolizers.
  Pharmacogenetic- Guided Metoprolol Management: A best practice advisory will be integrated into institutional clinical decision support systems for metoprolol dosing based on metabolic status of each patient.

SUMMARY:
Metoprolol is frequently administered to cardiac surgery patients to reduce the incidence of postoperative atrial fibrillation (PoAF). Metoprolol is metabolized by the enzyme CYP2D6, which is known to have many mutations that could influence a patient's ability to metabolize the drug. In this prospective clinical trial, the investigators will determine the genotype of CYP2D6 for patients undergoing cardiac surgery, provide an altered dosing recommendation for metoprolol, then report the relative effectiveness in managing PoAF for each pharmacogenetic- guided dosing category. The investigators will also explore the effects of personalized metoprolol dosing recommendations on outcomes in hospital length of stay, cost, and provider participation.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Scheduled for surgical procedure (coronary artery bypass graft and/or valve repair/replacement) at Vanderbilt University Medical Center

Exclusion Criteria:

* History of allergic reactions or contraindications to beta-blockers
* Patients with persistent atrial fibrillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2022-11-20 (Actual)

PRIMARY OUTCOMES:
Incidence of post-operative atrial fibrillation | From the end of anesthesia up to hospital discharge; usually 3-4 days
  Incidence of post-operative atrial fibrillation measured with post-operative electrocardiogram or rhythm strip, or at least two of the following: documentation in the progress notes, nursing notes, discharge summary, and change in medication.

SECONDARY OUTCOMES:
Rate of genome tailored prescription changes | From the end of anesthesia up to hospital discharge; usually 3-4 days
  Rate of genome tailored prescription changes as measured by the proportion of patients in whom metoprolol prescription is based on CYP2D6 metabolizer status.
Length of hospital stay | From end of surgery to hospital discharge; usually 3-4 days
  Length of hospital stay (in days) after surgery
Overall cost of treatment | From end of surgery to hospital discharge; usually 3-4 days
Cost of interventions to control or treat post-operative atrial fibrillation | From end of anesthesia to hospital discharge; usually 3-4 days
Incidence of adverse drug events | From end of anesthesia to hospital discharge; usually 3-4 days
Proportion of clinical decision support tool recommendations that were acknowledged and accepted by provider | From end of anesthesia to hospital discharge; usually 3-4 days
Proportion of clinical decision support tool recommendations that were acknowledged but ignored by the provider. | From end of anesthesia to hospital discharge; usually 3-4 days
Reasons for non-adherence to recommendations | From end of anesthesia to hospital discharge; usually 3-4 days
  Reasons for non-adherence to recommendations; prepopulated choices including 1. clinically inappropriate recommendation 2. provider preference 3. Other (free text option).

CONTACTS AND LOCATIONS:
Overall Officials: Miklos Kertai, MD. PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Staben R, Vnencak-Jones CL, Shi Y, Shotwell MS, Absi T, Shah AS, Wanderer JP, Beller M, Kertai MD. Preemptive Pharmacogenetic-Guided Metoprolol Management for Postoperative Atrial Fibrillation in Cardiac Surgery: The Preemptive Pharmacogenetic-Guided Metoprolol Management for Atrial Fibrillation in Cardiac Surgery Pilot Trial. J Cardiothorac Vasc Anesth. 2023 Oct;37(10):1974-1982. doi: 10.1053/j.jvca.2023.06.017. Epub 2023 Jun 14. PMID 37407326

DOCUMENTS (1):
  • Informed Consent Form (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/27/NCT03943927/ICF_000.pdf